CLINICAL TRIAL: NCT06997003
Title: Evaluation of a New Customized Corneal Treatment for Laser Refractive Vision Correction Using the TENEO™ 317 Model 2
Brief Title: Evaluation of a New Laser Refractive Vision Correction Using the TENEO™ 317 Model 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb GmbH (Industry)
Responsible Party: Sponsor
Organization: Bausch & Lomb Incorporated (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-LC04-TENOCT-6401
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hyperopia and Myopia
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyperopic eyes and anterior treatment mode (Experimental)
  Interventions: Device: Anterior treatment mode
- Myopic eyes and anterior treatment mode (Experimental)
  Interventions: Device: Anterior treatment mode
- Myopic eyes and total treatment mode (Experimental)
  Interventions: Device: Total treatment mode

INTERVENTIONS:
Device: Anterior treatment mode — Laser-in-situ-Keratomileusis (LASIK) surgery using OCTAVIUS treatment
  Arms: Hyperopic eyes and anterior treatment mode
Device: Anterior treatment mode — Laser-in-situ-Keratomileusis (LASIK) surgery using OCTAVIUS treatment
  Arms: Myopic eyes and anterior treatment mode
Device: Total treatment mode — Laser-in-situ-Keratomileusis (LASIK) surgery using OCTAVIUS treatment
  Arms: Myopic eyes and total treatment mode

SUMMARY:
Prospective, post market clinical follow up study with a three months postoperative follow up to evaluate the visual and refractive outcomes of OCTAVIUS treatment when used as intended.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects already scheduled for bilateral refractive laser surgery targeting emmetropia (attempted MRSE is between and including -0.50 D and +0.50 D).
2. Minimum 18 years of age.
3. Have read, understood, and signed an informed consent form (ICF).
4. Have a stable refraction (i.e., a change of ≤ 0.50 D in sphere and cylinder) for both eyes as judged by the investigator.
5. Have less than 0.75 D spherical equivalent (SE) difference between cycloplegic and manifest refractions at preoperative visit for both eyes.
6. Study group 1 only: Have hyperopic refractive error with or without astigmatism; sphere between 0.00 D and 4.00 D, cylinder between 0.00 D and 3.00 D for both eyes; with a spherical equivalent (SE) between 0.50 D and 5.50 D for both eyes.
7. Study groups 2 and 3 only: Have myopic refractive error with or without astigmatism; sphere between -8.00 D and 0.00 D, cylinder between 0.00 D and -4.00 D for both eyes; with a spherical equivalent (SE) between -10.00 D and -1.00 D for both eyes.
8. Have CDVA of 20/25 (logMAR 0.1) or better in both eyes
9. Have normal corneal topography as determined by the Investigator for both eyes.
10. Have discontinued use of contact lenses for at least 2 weeks (for hard lenses) or 3 days (for soft lenses) prior to the pre-operative examination, and through the day of surgery.
11. All contact lens wearers must demonstrate a stable refraction (within ± 0.50 D), as determined by MRSE, on two consecutive examinations at least 1 week apart, in both eyes and the axis of cylinder should not differ by more than 15 degrees from the baseline cycloplegic refraction for both eyes.
12. Have the ability to lie flat without difficulty.
13. Are willing and able to comply with the schedule for all post-surgery follow-up visits.

Exclusion Criteria:

1. Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns residual stroma thickness in any eye.
2. Tear Break-Up time (TBUT) <8 s in any eye.
3. Mesopic pupil size larger than the optical zone of the planned treatment for any eye.
4. History or evidence of active or inactive of corneal disease or infection in either eye (e.g., herpes simplex keratitis, herpes zoster keratitis, recurrent erosion syndrome, corneal dystrophy, etc.).
5. Central corneal scars affecting visual acuity or unstable keratometry with irregular mires in any eye.
6. Irregular astigmatism in any eye.
7. Keratoconus or suspicion of keratoconus (sub-clinical, forme fruste), corneal dystrophy in any eye.
8. Previous intraocular or corneal surgery in either eye that might confound the outcome of the study or increase the risk to the subject.
9. Ocular muscle disorder including a strabismus or nystagmus, or other disorder affecting fixation in any eye.
10. Evidence of retinal vascular disease in any eye.
11. History or evidence glaucoma or glaucoma suspect in any eye.
12. Acute or chronic disease or illness that would increase the operative risk, likely affect the wound healing or confound the outcomes of the study (e.g. immuno-compromised, connective tissue disease, clinically significant atopic disease, diabetes, etc.).
13. Use chronic systemic medications that may confound the outcome of the study or increase the risk to the subject, including, but not limited to steroids, antimetabolites, etc.;
14. Take medications contraindicated with LASIK such as isotretinoin (Accutane) or amiodarone hydrochloride (Cordarone).
15. Known sensitivity to medications used for standard LASIK treatment.
16. Females of childbearing potential (those who are not surgically sterilized or not postmenopausal for at least 12 months) if they meet one of the following conditions: Pregnant, lactating or unwilling to use effective birth control over the course of the study.
17. Concurrent or previous (within 30 days) participation in another drug or device investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of eyes that achieve a Uncorrected Distance Visual Acuity of 20/40 or better | Assessed for approximately 90 days
Percentage of participants with binocular Uncorrected Distance Visual Acuity of 20/40 or better | Assessed for approximately 90 days
Percentage of eyes that achieve predictability (attempted versus achieved) of Manifest Refraction Spherical Equivalent (MRSE) within ± 0.50 D | Assessed for approximately 90 days
Percentage of eyes that achieve predictability (attempted versus achieved) of Manifest Refraction Spherical Equivalent (MRSE) within ± 1.00 D | Assessed for approximately 90 days

SECONDARY OUTCOMES:
Preservation of Corrected Distance Visual Acuity (CDVA) | Assessed for approximately 90 days
  Percentage of eyes with CDVA worse than 20/40 at postoperative visit 3 if 20/20 or better preoperatively
Preservation of Corrected Distance Visual Acuity (CDVA) | Assessed for approximately 90 days
  Percentage of eyes with CDVA loss > 2 lines (> 10 letters ETDRS scale) at visit 3
Induced Manifest Refraction Astigmatism | Assessed for approximately 90 days
  Percentage of eyes that have a magnitude of postoperative manifest refractive astigmatism that increases from baseline cylinder by > 2.00 D at postoperative visit 3
Incidence of Adverse Events | Assessed from 0-90 days
  Percentage of eyes with treatment emergent adverse events occurred per event type

CONTACTS AND LOCATIONS:
Overall Officials: Natasa Orlic-Pleyer, Study Director — Bausch & Lomb GmbH
Locations (1):
- Site 01, Zlín, Czech Republic, Czechia